CLINICAL TRIAL: NCT04959539
Title: Endoscopic Transcanal Tympanoplasty With Attico-antrostomy Versus Endoscopic-assisted Canal Wall up Mastoidectomy in Management of Localized Cholesteatoma: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha A.Elkholy, Principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS/17.05.161
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Cholesteatoma
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic transcanal tympanoplasty with attico-antrostomy (Active Comparator)
  Interventions: Procedure: endoscopic transcanal tympanoplasty with attico-antrostomy
- endoscopic assisted canal wall up mastoidectomy (Active Comparator)
  Interventions: Procedure: endoscopic assisted canal wall up mastoidectomy

INTERVENTIONS:
Procedure: endoscopic transcanal tympanoplasty with attico-antrostomy — Transcanal approach followed by atticotomy to remove the attic cholesteatoma sac
  Arms: endoscopic transcanal tympanoplasty with attico-antrostomy
Procedure: endoscopic assisted canal wall up mastoidectomy — traditional canal wall up mastoidectomy followed by endoscopic evaluation of the attic to exclude any remnant cholesteatoma
  Arms: endoscopic assisted canal wall up mastoidectomy

SUMMARY:
the main objective of the study is to compare endoscopic transcanal tympanoplasty with attico-antrostomy with endoscopic assisted canal wall up mastoidectomy in treatment of limited attic cholesteatoma.

ELIGIBILITY:
Inclusion Criteria:

* Cases of cholesteatoma limited to the middle ear and/or attic but not extending beyond the posterior end of the lateral semicircular canal (LSCC) proved radiologically with computed tomography (CT) scan

Exclusion Criteria:

* Cases in which cholesteatoma extended beyond the attic were excluded as being potentially beyond the limits of the TEES approach

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
eradication of attic cholesteatoma | 6 months postoperative
  number of participants with no recurrence documented by second look surgery or MRI diffusion

CONTACTS AND LOCATIONS:
Locations (1):
- ORL-HNS department,Mansoura University Hospital, Faculty of Medicine, Mansoura University, Al Mansurah, ElDakahlia, Egypt

REFERENCES:
- [Derived] Moneir W, Hemdan A, El-Kholy NA, El-Kotb M, El-Okda M. Endoscopic transcanal attico-antrostomy versus endoscopic-assisted canal wall up mastoidectomy in management of localized cholesteatoma: a randomized clinical trial. Eur Arch Otorhinolaryngol. 2022 Sep;279(9):4371-4378. doi: 10.1007/s00405-021-07200-x. Epub 2021 Dec 1. PMID 34851451